CLINICAL TRIAL: NCT04829019
Title: A Randomised Controlled Trial to Investigate the Neurocognition in EGFR-mutant Advanced Non-small Cell Lung Cancer Patients With Symptomatic Brain Metastases Treated With Osimertinib or Osimertinib Plus Whole-brain Irradiation (WBI)
Brief Title: Neurocognition in NSCLC Patients Treated With Osimertinib or Osimertinib + WBI
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Li Zhang, MD, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESR-18-14285
Record Dates: First submitted 2021-03-31; First posted 2021-04-02 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2021-03

CONDITIONS: Neurocognitive
MeSH Terms: interventions — osimertinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- whole-brain irradiation (WBI) plus Osimertinib (Active Comparator): Osimertinib plus WBI, with Osimertinib at a dose of 80 mg once per day.
  Interventions: Radiation: Osimertinib and whole-brain irradiation
- Osimertinib (Active Comparator): Osimertinib with WBI sequential therapy, with Osimertinib at a dose of 80 mg once per day.
  Interventions: Drug: Osimertinib

INTERVENTIONS:
Radiation: Osimertinib and whole-brain irradiation — Osimertinib at a dose of 80 mg once per day, and WBI
  Arms: whole-brain irradiation (WBI) plus Osimertinib
Drug: Osimertinib — Osimertinib at a dose of 80 mg once per day, until unacceptable adverse events or disease progression occurred. WBI could be given to patients in experimental arm at any time base on investigator's decision after treatment initiated.
  Arms: Osimertinib

SUMMARY:
This is a prospective, randomised, positive-controlled, study to assess the neurocognitive function of upfront Osimertinib compared to whole-brain irradiation (WBI) plus Osimertinib in EGFR-mutant (Ex 19Del and L858R) NSCLC patients with symptomatic brain metastases, as well as the efficacy and safety.

DETAILED DESCRIPTION:
Account for patients with wild type EGFR, sample attrition , incidence rate of symptomatic brain metastasis(10%) and any other reasons for screen failure rate(50%), it is esimated that 88 patients will be randomized from 5 sites. Patients will be randomized 1:1, the experimental arm is upfront Osimertinib with WBI sequential therapy, while the control arm is Osimertinib plus WBI. Osimertinib at a dose of 80 mg once per day, until unacceptable adverse events or disease progression occurred. WBI could be given to patients in experimental arm at any time base on investigator's decision after treatment initiated. Patients will be stratifed at randomization by GPA score (3.5-4 vs <3.5) and the mutation type (Ex19Del / L858R). Patients will undergo the neurocognition, efficacy and safety assessments at baseline, and every 8 weeks until treatment is completed or discontinued. About time to brain metastases symptoms deterioration, the assessment was repeated in the first week (on site), second week (through telephone) and fourth week (on site). The rest assessment will be as well as other evaluations repeated every 8 weeks. To evaluate the correlation and predictive or prognostic value between gene dynamic changes and clinical efficacy, the tissue, plasma and cerebrospinal fluid (CSF) samples will be collected at baseline. CSF will be collected in patients with intracranial progression. Plasma will be collected in all the patients at disease progression, while tissue is optional. Also, plasma will be collected at week 8(first evaluation of efficacy).

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures
2. Male or female, aged at least 18 years
3. Eastern Cooperative Oncology Group (ECOG) performance-status score of 0 or 1
4. Life expectancy of at least 3 months
5. Histologically or cytologically documented metastatic NSCLC, which are not amenable to curative surgery or radiotherapy, patients must be classified as stage IIIB-IV. Staging will be according to the TNM staging system for lung cancer (8th edition)
6. Histologically documented that with sensitizing EGFR mutations(either L858R or Exon19del)
7. symptomatic brain metastasis, with at least three metastatic lesions in the brain which need WBI based on investigator's decision. Symptom score 1-6 point.(notes: Symptomatic definition: Symptoms without acute intervention or hospitalization, symptoms including but not limited in headache, nausea, dizziness, and sensory disturbance, but without hospitalization or medical emergency.)
8. HVLT-R score 15 point (Notes: this number is based on the data in a study in Chinese population)
9. At least 1 measurable lesion in the brain according to RECIST 1.1; At least one lesion, not previously irradiated, that can be accurately measured at baseline as ≥ 10 mm in the longest diameter with computed tomography (CT) or magnetic resonance imaging (MRI).
10. No previous treatment with EGFR-TKI or other systemic treatment, as well as radiotherapy for brain metastases.
11. Female subjects should be using highly effective contraceptive measures, and must have a negative pregnancy test and not be breast-feeding prior to start of dosing if of child-bearing potential, or must have evidence of non-child-bearing potential by fulfilling one of the following criteria at screening:

    * Post-menopausal defined as aged more than 50 years and amenorrheic for at least 12 months following cessation of all exogenous hormonal treatments
    * Women under 50 years old would be considered postmenopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and with LH and FSH levels in the post-menopausal range for the institution
    * Documentation of irreversible surgical sterilisation by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation Further information in Appendix E(Definition of Women of Childbearing Potential and Acceptable Contraceptive Methods)
12. Male subjects should be willing to agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures and agreement to refrain from donating sperm, as defined below: a. With female partners of childbearing potential or pregnant female partners, men must remain abstinent or use a condom during the treatment period and for at least 4 months after the last dose of Osimertinib. b. Men must refrain from donating sperm during this same period

Exclusion Criteria:

1. Involvement in the planning and/or conduct of the study (applies to both Investigator staff and/or staff at the study site)
2. Previous randomisation in the present study or previous treatment with osimertinib
3. Leptomeningeal met alone or synchronously is not allowed
4. History of hypersensitivity to active or inactive excipients of Osimertinib or drugs with similar chemical structure or class to Osimertinib
5. For patients, inability to collect plasma, CSF and tissue at baseline
6. Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension and active bleeding diatheses, which in the investigator's opinion makes it undesirable for the patient to participate in the trial or which would jeopardise compliance with the protocol, or active infection including hepatitis B, hepatitis C and human immunodeficiency virus (HIV). Screening for chronic conditions is not required.
7. Currently receiving (or unable to stop use prior to receiving the first dose of study treatment) medications or herbal supplements known to be strong inducers of CYP3A4 (at least 3 week prior) (Appendix D). All patients must try to avoid concomitant use of any medications, herbal supplements and/or ingestion of foods with known inducer effects on CYP3A4.
8. Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product or previous significant bowel resection that would preclude adequate absorption of osimertinib.
9. Any of the following cardiac criteria:

   * Mean resting corrected QT interval (QTc) > 470 msec obtained from 3 electrocardiograms (ECGs), using the screening clinic ECG machine derived QTc value (Note: patients with congenital long QT syndrome (CLQTS) are excluded from this study.)
   * Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG e.g. complete left bundle branch block, third degree heart block and second degree heart block.
   * Patient with any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, electrolyte abnormalities (including: Serum/plasma potassium < LLN; Serum/plasma magnesium < LLN; Serum/plasma calcium < LLN) , congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age in first degree relatives or any concomitant medication known to prolong the QT interval and cause Torsades de Pointes
10. Past medical history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis which required steroid treatment, or any evidence of clinically active interstitial lung disease.
11. Inadequate bone marrow reserve or organ function (as demonstrated by any of the following laboratory values:

    * Absolute neutrophil count <1.5 x 109/L;
    * Platelet count <100 x 109/L;
    * Haemoglobin <90 g/L;
    * Alanine aminotransferase >2.5 x ULN if no demonstrable liver metastases or >5 times ULN in the presence of liver metastases;
    * Aspartate aminotransferase >2.5 x ULN if no demonstrable liver metastases or >5 times ULN in the presence of liver metastases;
    * Total bilirubin >1.5 x ULN if no liver metastases or >3 x ULN in the presence of documented Gilbert's Syndrome [unconjugated hyperbilirubinaemia] or liver metastases;
    * Serum creatinine >1.5 x ULN concurrent with creatinine clearance <50 mL/min [measured or calculated by Cockcroft and Gault equation]
12. Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements.
13. Women who are pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2021-04-07 (Estimated); Primary Completion 2024-04-01 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
neurocognitive function (HVLT-R) | at 4 months
  measured as a significant deterioration (5-point drop compared with baseline) in Hopkins Verbal Learning Test-Revised (HVLT-R) total recall at 4 months

SECONDARY OUTCOMES:
intracranial progression-free survival | assessed up to 36 months
  defined as the time from randomization to the date of intracranial disease progression
progression-free survival | assessed up to 36 months
  defined as the time from randomization to the date of first documentary disease progression
intracranial overall response rate | assessed up to 60 months
  percentage of participants with objective response in brain metastasis
overall response rate | assessed up to 60 months
  percentage of participants with objective response
intracranial disease control rate | assessed up to 60 months
  percentage of participants with disease control in brain metastasis
disease control rate | assessed up to 60 months
  percentage of participants with disease control
intracranial Duration of Response | assessed up to 60 months
  defined as the time from randomization to the date of first documentary PR or CR in brain metastasis
Duration of Response | assessed up to 60 months
  defined as the time from randomization to the date of first documentary PR or CR
Time to initiate WBI | assessed up to 36 months
  defined as the time from randomization to the date of initiate WBI

OTHER OUTCOMES:
Health Related Quality of Life (HRQoL) | assessed up to 60 months
  Questionnaire consisting of 30 items measuring subjects general cancer symptoms and functioning
disease-related symptoms | assessed up to 60 months
  A complementary questionnaire measuring lung cancer symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Ting Zhang, Principal Investigator — Sun Yat-sen University
Locations (1):
- Department of Medical Oncology, Cancer Center of Sun Yat-Sen University, Guangzhou, Guangdong, China